CLINICAL TRIAL: NCT04824443
Title: Exercise Therapy in Cancer Patients Hospitalized for COVID-19: A Digitized Clinical Trial
Brief Title: Exercise Therapy in Cancer Patients Who Are Recovering From COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-101
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Covid19; Coronavirus; Cancer
Keywords: Covid19; Coronavirus; Cancer; Exercise; 21-101; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants who were hospitalized for COVID-19 (Experimental): Participants will be post-cancer treatment patients who were hospitalized for COVID-19.
  Interventions: Other: Aerobic Exercise Therapy

INTERVENTIONS:
Other: Aerobic Exercise Therapy — Aerobic Exercise Therapy/AT will consist of 30 weeks of treadmill walking sessions. AT will consist of supervised, individualized walking delivered up to 6 times weekly (over a 7-day period) to achieve a cumulative total duration ranging from 90 mins/wk up to 375 mins/wk following a non-linear dosing schedule. The planned dose and scheduling of AT will be continually altered and progressed in conjunction with appropriate rest/recovery sessions across the entire intervention period (i.e., non-linear periodized schedule).
  Other Names: AT

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a 30-week aerobic exercise therapy program in cancer patients recovering from COVID-19. The study will look at whether the aerobic exercise therapy causes few or mild side effects in participants. Aerobic exercise is physical activity that uses the large muscle groups (muscles in your legs, buttocks, back, and chest) and can be performed for several minutes at a time. The aerobic exercise therapy being used in this study will be a walking program that will be adjusted so it matches participant fitness levels (how much exercise you can handle).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Previously admitted to a hospital for Covid-19
* Discharged from hospital for at least 30 days
* Previously treated for cancer at MSK
* Interval of ≥ 12 months but ≤ 10 years following completion of primary non-hormonal anti-cancer therapy (current endocrine therapy and maintenance therapy allowed)
* Space to house a treadmill at personal residence
* Cleared for exercise participation as per screening clearance via the Physical Activity Readiness Questionnaire (PAR-Q+)
* Performing less than 90 minutes of structured moderate-intensity or strenuous-intensity exercise per week, as evaluation by self-report
* If a female of child-bearing potential, must not be pregnant or planning to become pregnant during the study.

  * Women <50 years old who are of child-bearing potential must have a negative pregnancy test within 14 days of enrollment.

Exclusion Criteria:

* Currently receiving home oxygen after discharge
* Enrollment onto any other interventional investigational study
* Current treatment for any other diagnosis of invasive cancer of any kind
* Distant metastatic malignancy of any kind
* Receiving non-hormonal anticancer therapy
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Frequency of serious adverse events during study-related assessments | 30 weeks
  Safety will be evaluated by the frequency of serious (i.e., life-threatening, hospitalization, significant incapacity, important medical events) adverse events during study-related assessments and exercise sessions according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Scott, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Scott JM, Qiu Z, Rahman J, Moskowitz CS, Michalski MG, Lehman S, Lee CP, Harrison J, Yu AF, Marouf A, Vardhana S, Boutros PC, Jones LW. Case Report: Decentralized trial of tolerability-adapted exercise therapy after severe Covid-19. Front Immunol. 2025 Apr 3;16:1529385. doi: 10.3389/fimmu.2025.1529385. eCollection 2025. PMID 40248705
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org